CLINICAL TRIAL: NCT04491656
Title: Evaluating Clinical Outcomes for Determining the Optimal Delay to Skin Incision Under WALANT: a Prospective Series of 34 Patients From a Low Resource Tertiary Setting
Brief Title: Evaluating Clinical Outcomes for Determining the Optimal Delay to Skin Incision Under WALANT
Acronym: WALANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Avenue Medical Center, Philippines (Other Government)
Responsible Party: Principal Investigator, Alvin A. Hernandez, Principal Investigator, East Avenue Medical Center, Philippines
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EAMC IERB 2020 - 03
Record Dates: First submitted 2020-07-23; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Hand Surgery; Orthopedic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7 minutes group (Active Comparator): surgeries performed with this group would wait 7 minutes after lidocaine+epinephrine injection prior to skin incision
  Interventions: Other: WALANT Technique
- 30 minutes group (Active Comparator): surgeries performed with this group would wait 30 minutes after lidocaine+epinephrine injection prior to skin incision
  Interventions: Other: WALANT Technique

INTERVENTIONS:
Other: WALANT Technique — A technique commonly used in hand surgeries where the combination of lidocaine and epinephrine is used for local blood control, thus performing the procedure without a tourniquet

SUMMARY:
Further studies are needed to establish the effects of WALANT in performing most common hand surgeries, in relation to its clinical outcomes and intraoperative blood loss. Therefore, this study aims to identify the best interval time to perform elective hand surgeries using WALANT technique, document clinical outcomes and identify potential complications

DETAILED DESCRIPTION:
To propose the optimal time delay from the injection to skin incision for most WALANT surgeries of the hand or wrist by analyzing not only intraoperative blood loss, but also postoperative pain scores and complication rates

To determine if there is a difference between performing the WALANT technique with a waiting interval of 7 minutes as compared to 30 minutes prior to incision in relation to blood loss, pain scores, and complications.

Initiate the use of WALANT technique and its application in practice of Orthopaedic Residents in East Avenue Medical Center

ELIGIBILITY:
Inclusion Criteria:

1. . Signed Consent Form
2. Elective Hand Surgeries
3. Minor Hand Surgeries
4. Adult Male/Female ages 18 and above
5. Multiply injured

Exclusion Criteria:

1. No Consent
2. Multiply injured patient
3. Traumatic Hand Injuries
4. Known allergic reaction to either Epinephrine or Lidocaine.
5. Known heart condition
6. Patients on anticoagulants
7. Patients diagnosed with bleeding disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
VRS Score | 24 weeks
  Verbal Rating Scale
  1. 0 for no pain
  2. 1 for mild pain
  3. 2 for moderate pain
  4. 3 for severe pain
  5. 4 for very severe pain

SECONDARY OUTCOMES:
Blood Loss | 24 weeks
  Blood loss estimation using Gauze Visual Analogue Scale by Algadiem et.al.

OTHER OUTCOMES:
Complications | 24 weeks
  Complications which may occur during the course of treatment and subsequent follow up of the patients which includes: wound complications, infection, stiffness, pain

CONTACTS AND LOCATIONS:
Overall Officials: Mamer S. Rosario, MD, Study Chair — East Avenue Medical Center, Department of Orthopedics
Locations (1):
- East Avenue Medical Center; Department of Orthopedics, Quezon City, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Patient DATA will remain anonymous during the study and to be coded. Outcome measures for all participants will be documented
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: August 2020